CLINICAL TRIAL: NCT01444495
Title: Randomized Clinical Trial on Preoperative Radiotherapy 25 Gy in Rectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Radoslaw Pach, MD, PhD, Assisstant Professor, Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Cracow Rectal Cancer Trial
Record Dates: First submitted 2011-09-29; First posted 2011-09-30 (Estimated); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Rectal Cancer
Keywords: rectal cancer; radiotherapy; overall survival; recurrence rate; downstaging
MeSH Terms: conditions — Rectal Neoplasms | interventions — Neoadjuvant Therapy; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short time interval (Active Comparator): Patients operated on 7-10 days after completing preoperative radiotherapy 5x5Gy.
  Interventions: Radiation: Preoperative radiotherapy; Procedure: Surgery
- Long time interval (Experimental): Patients operated on 4-5 weeks after completing preoperative radiotherapy 5x5Gy.
  Interventions: Radiation: Preoperative radiotherapy; Procedure: Surgery

INTERVENTIONS:
Radiation: Preoperative radiotherapy — Preoperative radiotherapy 5x5 Gy (total dose of 25 Gy)
  Other Names: Neoadjuvant radiotherapy
Procedure: Surgery — Total mesorectal excision of rectal cancer
  Other Names: Operative treatment

SUMMARY:
The purpose of this study is to establish the influence of time-interval between preoperative hyperfractionated radiotherapy (5x5 Gy) and surgery on long term overall survival (5 years), local and distant recurrence rate, downstaging rate, sphincter saving procedures, radical resection rate (R0) in patients with locally advanced rectal cancer operated on according to TME technique. In particular 3D endosonography and 3rd generation ultrasonic contrast agents are evaluated to assess response to radiotherapy.

DETAILED DESCRIPTION:
The treatment group comprises patients with locally advanced rectal cancer who were operated on in the 1st Department of General Surgery, Jagiellonian University, Cracow. The data on survival has been systematically collected using national census registry. Patients are qualified to preoperative radiotherapy 5x5 Gy and then randomly assigned to subgroups with different time interval between radiotherapy and surgery: one subgroup consists of patients operated on 7-10 days after the end of irradiation, the second subgroup consists of patients operated on after 4-5 weeks. Both should be homogenous in sex, age, cancer stage and localization, distal and circumferential resection margins, number of resected lymph nodes. 3D endorectal ultrasound and endorectal ultrasound with SonoVue are performed to assess the tumor before and after preoperative radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed rectal cancer
* tumor localised in middle or lower rectum
* age > 18 years
* locally advanced cancer

Exclusion Criteria:

* previous pelvis radiotherapy
* lack of patient's consent
* lack of possibility to begin radiotherapy during 14 days after inclusion to the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 1999-01; Primary Completion 2008-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
local and systemic recurrence rate | 5 years
  Rate of local and sytemic recurrences in patients included to the protocol.

SECONDARY OUTCOMES:
radical resections rate (R0) | 1 month
  Rate of R0, R1 and R2 procedures according to Hermanek.
sphincter saving (sparing) procedures | 1 month
  Rate of sphincter saving operations in both arms.
overall survival | 5 years
  Overall survival and disease specific survival at 5 years follow-up
downstaging of rectal cancer | 1 month
  Downstaging of the rectal cancer after preoprearite radiotherapy - assessed by comparison of preoperative ERUS, 3D ERUS, contrast enhanced ERUS and postoperative histologic staging

CONTACTS AND LOCATIONS:
Overall Officials: Jan Kulig, Prof., Study Chair — First Department of General Surgery, Jagiellonian University; Radoslaw Pach, Ph.D., Principal Investigator — First Department of General Surgery, Jagiellonian University
Locations (1):
- First Department of Surgery, Krakow, Malopolska, Poland

REFERENCES:
- [Result] Pach R, Kulig J, Richter P, Gach T, Szura M, Kowalska T. Randomized clinical trial on preoperative radiotherapy 25 Gy in rectal cancer--treatment results at 5-year follow-up. Langenbecks Arch Surg. 2012 Jun;397(5):801-7. doi: 10.1007/s00423-011-0890-8. Epub 2011 Dec 15. PMID 22170083
- [Result] Pach R, Kulig J, Richter P, Gach T, Szura M, Kowalska T. Erratum to: Randomized clinical trial on preoperative radiotherapy 25 Gy in rectal cancer-treatment results at 5 year follow-up. Langenbecks Arch Surg. 2019 Sep;404(Suppl 1):19-20. doi: 10.1007/s00423-012-0940-x. No abstract available. PMID 22398435
- [Result] Pach R, Sierzega M, Szczepanik A, Popiela T, Richter P. Preoperative radiotherapy 5 x 5 Gy and short versus long interval between surgery for resectable rectal cancer: 10-Year follow-up of the randomised controlled trial. Radiother Oncol. 2021 Nov;164:268-274. doi: 10.1016/j.radonc.2021.10.006. Epub 2021 Oct 13. PMID 34653526
- [Result] Pach R, Richter P, Sierzega M, Papp N, Szczepanik A. Preoperative Short-Course Radiotherapy and Surgery versus Surgery Alone for Patients with Rectal Cancer: A Propensity Score-Matched Analysis at 18-Year Follow-Up. Biomedicines. 2021 Jun 24;9(7):725. doi: 10.3390/biomedicines9070725. PMID 34202691
- [Result] Pach R, Szczepanik AM, Sierzega M, Daniluk M, Richter P. Prognostic value of lymph node ratio in resectable rectal cancer after preoperative short-course radiotherapy-results from randomized clinical trial. Langenbecks Arch Surg. 2022 Nov;407(7):2969-2980. doi: 10.1007/s00423-022-02603-8. Epub 2022 Jul 4. PMID 35788774